CLINICAL TRIAL: NCT00458120
Title: Evaluation of the Safety and Immunogenicity of Heterologous Dengue Vaccine Administration in Dengue Immune Individuals
Brief Title: Safety of and Immune Response to Two Different Dengue Virus Vaccines in Individuals Previously Immunized Against Dengue Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 227; WIRB Protocol Number 20070409
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; Dengue Vaccination
MeSH Terms: conditions — Severe Dengue; Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Participants previously vaccinated with rDEN4delta30 will receive one subcutaneous vaccination (10^3 dose of vaccine) of rDEN1delta30 vaccine into the deltoid region of either arm.
  Interventions: Biological: rDEN1delta30
- 2 (Experimental): Participants previously vaccinated with rDEN4delta30 will receive one subcutaneous vaccination (10^3 dose of vaccine) of rDEN2/4delta30(ME) into the deltoid region of either arm.
  Interventions: Biological: rDEN2/4delta30(ME)
- 3 (Experimental): Participants previously vaccinated with rDEN2/4delta30(ME) will receive one subcutaneous vaccination (10^3 dose of vaccine) of rDEN1delta30 vaccine into the deltoid region of either arm.
  Interventions: Biological: rDEN1delta30
- 4 (Experimental): Participants previously vaccinated with rDEN1delta30 will receive one subcutaneous vaccination (10^3 dose of vaccine) of rDEN2/4delta30(ME) vaccine into the deltoid region of either arm.
  Interventions: Biological: rDEN2/4delta30(ME)
- 5 (Placebo Comparator): One subcutaneous vaccination with placebo into the deltoid region of either arm.
  Interventions: Biological: Placebo to rDEN1delta30 or rDEN2/4delta30(ME)

INTERVENTIONS:
Biological: rDEN1delta30 — Live attenuated 10^3 dose of rDEN1delta30 vaccine. Participants must have been previously vaccinated with rDEN4delta30 or rDEN2/4delta30(ME) vaccines.
  Arms: 1; 3
Biological: rDEN2/4delta30(ME) — Live attenuated 10^3 dose of rDEN2/4delta30(ME) vaccine. Participants must have been previously vaccinated with rDEN4delta30 or rDEN1delta30 vaccines.
  Arms: 2; 4
Biological: Placebo to rDEN1delta30 or rDEN2/4delta30(ME) — Placebo vaccines for rDEN1delta30 and rDEN2/4delta30(ME)
  Arms: 5

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in subtropical regions of the world. There are four different forms (serotypes) of dengue virus that can cause dengue fever. The purpose of this study is to determine the safety and immune response to a vaccine containing a particular dengue serotype when an individual has been previously vaccinated with a different dengue serotype.

DETAILED DESCRIPTION:
The World Health Organization estimates that dengue virus causes more than 50 million cases of dengue fever a year. Dengue virus infection is the leading cause of hospitalization and death in children of most tropical Asian countries. There are four different serotypes of dengue virus. Most cases of dengue hemorrhagic fever/dengue shock syndrome are caused by secondary infection with a dengue serotype different from the first serotype the individual was infected with. A vaccine that would be effective in preventing infection by multiple dengue serotypes is desirable. The purpose of this study is to determine the safety of and immune response to two different dengue virus vaccines in individuals who have been previously vaccinated against a different serotype.

This study will last at least 42 days. Participants will be recruited from a database of previous dengue vaccine recipients and will be stratified by the type of vaccine previously received. Participants assigned to Cohort 1 and Cohort 2 will have already been vaccinated with the rDEN4delta30 vaccine. Participants assigned to Cohort 3 will have already been vaccinated with the rDEN2/4delta30(ME) vaccine. Participants in Cohort 4 will have already been vaccinated with the rDEN1delta30 vaccine. Participants in Cohorts 1 and 3 will be randomly assigned to receive either the rDEN1delta30 vaccine or placebo. Participants in Cohorts 2 and 4 will be randomly assigned to receive either the rDEN2/4delta30(ME) vaccine or placebo.

Participants will receive their assigned vaccination on Day 0. Study visits will occur every other day until Day 16, and then at Days 21, 28, and 42. At each visit, blood collection, vital signs measurement, and a physical exam will occur. In addition, participants will be asked to monitor their temperature daily, 3 times a day, from Day 0 to Day 16. Patients will also be asked to enroll in an optional skin biopsy sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Previous vaccination with rDEN1delta30, rDEN2/4delta30(ME), OR rDEN4delta30 vaccine
* General good health
* Available for the duration of the study
* Willing to use accepted forms of contraception

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease by history, physical examination, or laboratory studies including urinalysis
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may interfere with the study
* Certain abnormal laboratory values
* Medical, work, or family problems as a result of alcohol or illegal drug use within 12 months of study entry
* History of severe allergy or anaphylaxis
* Severe asthma requiring an emergency room visit or hospitalization within 6 months of study entry
* HIV infected
* Hepatitis C virus infected
* Hepatitis B surface antibody positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs 30 days prior to study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Receipt of live vaccine within 4 weeks of study entry
* Receipt of killed vaccine within 2 weeks of study entry
* Absence of spleen
* Plan to travel to an area where dengue virus is common
* Any investigational product within 30 days of study entry
* Other condition that, in the opinion of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Number, severity, and seriousness of vaccine-related adverse events observed through active and passive surveillance | Throughout study
Neutralizing antibody to all four dengue serotypes | At Days 0, 28, and 42

SECONDARY OUTCOMES:
Assess the frequency, quantity, and duration of viremia in each vaccine cohort studied | Throughout study
To determine if cellular targets of vaccine infection, including peripheral blood mononuclear cells and skin, are different after heterologous infection of a second dengue virus vaccine of a different serotype | Throughout study
Compare the safety and immunogenicity between each heterologous dengue vaccine virus cohort | At study completion
Evaluate the immunopathological mechanism of heterologous vaccine virus associated rash in those volunteers who are willing to undergo skin biopsy | Throughout study
Characterize the antibody response after heterolouous vaccine infection | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Durbin AP, Whitehead SS, McArthur J, Perreault JR, Blaney JE Jr, Thumar B, Murphy BR, Karron RA. rDEN4delta30, a live attenuated dengue virus type 4 vaccine candidate, is safe, immunogenic, and highly infectious in healthy adult volunteers. J Infect Dis. 2005 Mar 1;191(5):710-8. doi: 10.1086/427780. Epub 2005 Jan 27. PMID 15688284
- [Background] Chaturvedi UC, Shrivastava R, Nagar R. Dengue vaccines: problems and prospects. Indian J Med Res. 2005 May;121(5):639-52. PMID 15937367
- [Background] Guzman MG, Mune M, Kouri G. Dengue vaccine: priorities and progress. Expert Rev Anti Infect Ther. 2004 Dec;2(6):895-911. doi: 10.1586/14789072.2.6.895. PMID 15566333
- [Derived] Durbin AP, Schmidt A, Elwood D, Wanionek KA, Lovchik J, Thumar B, Murphy BR, Whitehead SS. Heterotypic dengue infection with live attenuated monotypic dengue virus vaccines: implications for vaccination of populations in areas where dengue is endemic. J Infect Dis. 2011 Feb 1;203(3):327-34. doi: 10.1093/infdis/jiq059. Epub 2010 Dec 14. PMID 21208923